CLINICAL TRIAL: NCT00976872
Title: Supplementation of Omega-3 Fatty Acid Complex to Routine Statin Treatment Decreases Patients' Day-time Blood Pressure, Improves Inflammatory Status and Prohibits Platelet Aggregation
Brief Title: Omega 3 Action on Cardiovascular Risk Factors in Patients Treated With Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Keren Doenyas-barak, Assaf-HarofehMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: keren1
Record Dates: First submitted 2009-09-13; First posted 2009-09-15 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2009-09

CONDITIONS: Inflammation; Blood Pressure; Platelet Function; Endothelial Function
Keywords: omega 3; inflammation; augmentation index; endothelial function
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega-3 (Active Comparator): omega-3: 2 pills of Omega"950"®, Solgar, New Jersey, USA. Each pill contained 542mg of eicosapentaenoic acid, EPA, and 405mg of docosahexanoic acid, DHA
  Interventions: Drug: omega-3
- placebo (Placebo Comparator): hard gelatin capsule of Capsugel®, France, filled with 1ml of soya oil
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omega-3 — omega-3: 2 pills of Omega"950"®, Solgar, New Jersey, USA. Each pill contained 542mg of eicosapentaenoic acid, EPA, and 405mg of docosahexanoic acid, DHA
  Arms: omega-3
Drug: placebo — hard gelatin capsule of Capsugel®, France, filled with 1ml of soya oil
  Arms: placebo

SUMMARY:
Recent evidences showed beneficial effects of omega-3 fatty acids on cardiovascular morbidity and mortality.

Regular Omega-3 fatty acid consumption reduces cardiovascular mortality, ischemic heart disease and stroke mortality. There is probably no single mechanism of action that explains this beneficial effect; but possible mechanisms include reduce susceptibility of the heart to ventricular arrhythmia, antithrombogenic effect, reduce triglyceride level, promotion of nitric oxide-induced endothelial relaxation, and retard growth of atherosclerotic plaque.

The combination of satins and omega3 was proved to be better the any of the drugs alone in several studies.

The purpose of the study is to investigate several possible mechanisms that may explain the add on beneficial effect of omega-3 in hypercholesterolemic patients already treated with satins.

DETAILED DESCRIPTION:
Cardiovascular disease is a leading cause of death in the western world. HMG-co A Reductase (statins) stands in the first line of treatment of cardiovascular disease because of their direct effect on LDL and their pleotrophic effect (mainly anti-inflammatory).

Recent evidences showed beneficial effects of omega-3 fatty acids on cardiovascular morbidity and mortality

Regular Omega-3 fatty acid consumption reduces cardiovascular mortality , , ischemic heart disease and stroke mortality. There is probably no single mechanism of action that explains this beneficial effect; but possible mechanisms include reduce susceptibility of the heart to ventricular arrhythmia, antithrombogenic effect , reduce triglyceride level , promotion of nitric oxide-induced endothelial relaxation , , and retard growth of atherosclerotic plaque.

Statins have a proven survival benefit in patients with hypercholesterolemia by preventing both primary and secondary cardiovascular events . Statins also has beneficial effect on lipid profile (mainly LDL and less triglycerides), they reduce plaque growth and improves endothelial function.

Many studies have demonstrated the additive effect of the combination of statins and omega-3 fatty acids on lipid profile, as well as additive effect on inflammatory markers (IL-6 and CRP).

JELIS 3is a recent study that examined 19000 patients with hypercholesterolemia treated with statins. This study demonstrated 19% reduction in coronary events under statins and omega 3 co-treatment.

The purpose of the study is to investigate several possible mechanisms that may explain the add on beneficial effect of omega-3 in hypercholesterolemic patients already treated with satins.

Methods 80 patients age 30-70 with known dyslipidemia treated with statins will be enrolled at the research center in Asaf-Harofeh medical center.

All patients will pass an interview, physical examination, lipid profile, CBC; and glucose level at base line.

Exclusion criteria: thrombocytopenia, bleeding disorder, uncontrolled hypertension, LDL>160, uncontrolled diabetes mellitus, recent (3m) cardiovascular event, or omega-3 pretreatment.

During the first 3 weeks all the patients will receive placebo. After randomization 40 patients will receive Omega-3 (2 pills omega-950, Solgar, every day) for the next 5 months, 40 patients will receive placebo.

At baseline, after 3 weeks of placebo and after 6 weeks of omega-3 treatment, and after another 3 months, all patients will come to the research center and have interview, physical examination, lipid profile, including oxidized LDL. In order to learn about inflammation we will measure hsCRP, we will measure Isoprostane as a marker for oxidative stress,Lp-PLA2 will be measures in order to learn about plaque activity, Augmentation index will be measured to learn about arterial stiffness and central hypertension, platelet aggregation tests in a new method called cone and platelet analyzer will be measured. In every meeting a blood pressure recorder will measure 24h blood pressure.

Augmentation index:

Brachial blood pressure will be measured using a validated, manual oscillometric device .Patients were seated and rested for 5 minutes in a quiet room, after which time blood pressure will be measured over the brachial artery 3 times at 5-minute intervals. The mean of the last 2 measurements was recorded as representative of brachial blood pressure. After the last measurement, radial artery pressure waveforms of the same arm will be sampled over 10 seconds with a Millar tonometer (SPC-301, Millar Instruments) and calibrated to the average blood pressure. Waveforms were then processed with dedicated software (SphygmoCor version 7, AtCor). The integral system software will be used to calculate an averaged radial artery waveform and to derive a corresponding central aortic pressure waveform using a previously validated generalized transfer function. Aortic pressure waveforms will be subjected to further analysis by the SphygmoCor software to identify the time to the peak/shoulder of the first and second pressure wave components (T1, T2) during systole. The pressure at the peak/shoulder of the first component will be identified as P1 height (outgoing pressure wave), and the pressure difference between this point and the maximal pressure during systole ( P or augmentation) will be identified as the reflected pressure wave occurring during systole. Augmentation index (AIx), defined as the ratio of augmentation to central pulse pressure, is expressed as a percentage: AIx=( P/PP)x100, where P is pressure and PP is pulse pressure.

Cone and platelet analyser:

The CPA tests platelet activation in whole blood under flow conditions. 200 µL of citrated blood will be placed in polystyrene wells and circulated at a high shear rate (1875 s-1) for 2 minutes with a rotating Teflon cone. Wells will be washed with water, stained (May-Grünwald), and analyzed with an inverted-light microscope connected to an image analysis system. Results are expressed as the percentage of the well surface covered by platelets.

Isoprostane Isoprostane is a marker for oxidative stress. Isoprostane level is measured by EIA (Cayman Chemical Company)

Blood Pressure monitor:

Twenty-four-hour ABPM will be executed with Spacelabs 90207. The monitor was mounted on the nondominant arm between 8:00 AM and 10:00 AM and removed 24 hours later. Recordings were made every 20 minutes between 6:00 AM and midnight and every 30 minutes between midnight and 6:00 AM.

Patients will be classified as having normal awake BP if the corresponding value was <135-mm Hg systolic BP (SBP) and <85-mm Hg diastolic BP (DBP). Normal sleep BP was considered <120/70 mm Hg.20,21 The overall 24-hour normality definition was <125/80 mm Hg.22 The normal dip was defined separately for SBP and DBP as 10% reduction in BP during sleep compared with the awake period.23 Nondipping was defined as a decrease <10% but 0%. Dipping beyond 20% was considered "extreme," and sleep-related BP "rising" denoted negative dipping.

PLAC The PLAC Test is a blood test that measures the level of Lp-PLA2, an enzyme highly specific to vascular inflammation and implicated in the formation of rupture-prone plaque.

The PLAC Test is the only blood test cleared by the FDA to aid in assessing risk of both coronary heart disease and ischemic stroke associated with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* dyslipidemia controlled (LDL < 130)
* statin treatment
* triglycerides < 200
* informed consent

Exclusion Criteria:

* thrombocytopenia or bleeding tendency
* uncontrolled diabetes mellitus
* uncontrolled hypertension (systolic > 160 or diastolic > 100)
* omega 3 pretreatment
* recent acute coronary syndrome or cerebrovascular event (less than 3 months)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
augmentation index | 0, 3 weeks, 6 weeks, 20 weeks
  Each patient was seated in a quiet room, blood pressure was measured. Radial artery pressure waveform was sampled with a Millar tonometer (SPC-301, Millar Instruments) and calibrated to the average blood pressure. Waveforms were then processed using the specific software (SphygmoCor, version 7, AtCor). Integral system software was used for calculation of the averaged radial artery waveform and derivation of the corresponding central aortic pressure waveform, using a previously validated generalized transfer function.

SECONDARY OUTCOMES:
blood pressure (24 hours monitor) | 0, or 3 weeks, 6 weeks, 20 weeks
  Twenty-four-hour - ambulatory blood pressure monitoring was performed using the SpacelabsTM 90207 ambulatory blood pressure monitor (ABPM). The monitor was mounted on the non-dominant arm in the morning (8:00 AM to 10:00 AM) and removed following 24h. The recordings were registered every 20 minutes between 6:00 AM and midnight, and every 30 minutes between midnight and 6:00 AM. Based on these measurements, the mean values and the loads of blood pressure were calculated.
platelet function | 0, 3 weeks, 6 weeks, 20 weeks
  CPA method was applied for analyzing the capacity of platelets to aggregate and adhere in whole blood under flow conditions. In brief, 200 µL of citrated blood was placed into polystyrene wells and subjected to circulation at a high shear rate (1875 s-1) for 2 minutes with a rotating Teflon cone. The wells were then rinsed with water, stained by May-Grünwald dye and analyzed under inverted light microscope connected to an image analysis system.The results were expressed as percentages of the well surface covered by platelets and as the average size of the stained objects.
Isoprostane | 0, 3 weeks, 6 weeks, 20 weeks
  STAT-8-Isoprostane levels were assessed by a specific EIA kit (Cayman Chemicals, USA).
PAI-1, TNF-alpha, IL6 | 0, 3,6 and 20 weeks
  PAI-1, TNF-alpha and IL-6 were also measured by specific ELISAs (R &D, USA), according to the manufacturers' instructions.

CONTACTS AND LOCATIONS:
Overall Officials: shai efrati, Study Director — asaf-harofe medical center